CLINICAL TRIAL: NCT07215520
Title: A Double-blind, Randomized, Controlled, Phase 2a Study to Evaluate the Safety and Tolerability of a Newcastle Disease Virus-based Mucosal Vaccine (NDV-HXP-S-KP.2) Relative to an Approved Systemic mRNA Vaccine in Previously Vaccinated Adults
Brief Title: Safety and Tolerability of a Newcastle Disease Virus-Based Mucosal COVID-19 Vaccine in Previously Vaccinated Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CastleVax Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVX NDV-HXP-S-KP.2-2a
Record Dates: First submitted 2025-10-01; First posted 2025-10-10 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IN administration of study drug plus placebo via IM (Experimental): Nasal Administration of NDV-HXP-S-KP.2 and administration of placebo via Intramuscular Injection
  Interventions: Biological: NDV-HXP-S-KP.2
- IN administration of placebo plus COVID-19 vaccine via IM (Active Comparator): Nasal Administration of Placebo plus administration of COVID-19 mRNA vaccine via Intramuscular Injection
  Interventions: Biological: COVID-19 mRNA Vaccine

INTERVENTIONS:
Biological: NDV-HXP-S-KP.2 — Nasal Administration of a COVID-19 vaccine to compare against a commercially available mRNA vaccine
  Arms: IN administration of study drug plus placebo via IM
Biological: COVID-19 mRNA Vaccine — Used as a comparator to study vaccine
  Arms: IN administration of placebo plus COVID-19 vaccine via IM

SUMMARY:
A Double-blind, Randomized, Controlled, Phase 2a Study to Evaluate the Safety and Tolerability of a Newcastle Disease Virus-based Mucosal Vaccine (NDV-HXP-S-KP.2) Relative to an Approved Systemic mRNA Vaccine in Previously Vaccinated Adults

DETAILED DESCRIPTION:
This is a double-blind (supported by a double-dummy design), randomized, active comparator-controlled Phase 2a safety and tolerability study. The study will enroll approximately 200 previously COVID-19-vaccinated, male and nonpregnant female adult participants aged ≥18 years. Participants 18 through 64 years of age must have at least 1 underlying condition that puts them at high risk for severe outcomes from COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Is an adult 18 through 64 years of age at time of screening with at least 1 underlying condition that puts the participant at high risk for severe outcomes of COVID-19 per self-report OR is an adult ≥65 years of age at time of screening (with or without at least 1 underlying condition).
2. Has completed any WHO/FDA-authorized or approved primary COVID-19 vaccination series per self-report.
3. Has received last COVID-19 vaccine ≥6 months prior to study vaccination.
4. If a female of childbearing potential who is sexually active, agrees to use an adequate method of birth control from Screening through 90 days after study vaccination, and has used an adequate birth control method for at least 30 days prior to Screening. Sexually active male participants, unless the participant is sterile or otherwise unable to produce sperm, or has exclusively male sexual partners, must agree to abstinence or to use a barrier method (e.g., male condom) from vaccination through 90 days after study vaccination. Male participants must also agree to not donate sperm from vaccination through 90 days after study vaccination.
5. Is medically stable, as determined by the site investigator (based on review of health status, vital signs, medical history, and physical examination).
6. Agrees to not participate in any other SARS-CoV-2 infection prevention trial (vaccine, drug, biologic, pre-exposure prophylaxis [PrEP]) during participation in the study.
7. Willing and able to provide informed consent prior to initiation of study procedures.
8. Is available for all study visits, willing to participate in all study procedures, and not planning to relocate from the area for the duration of the study.

Exclusion Criteria:

1. Has an acute illness, as determined by the site investigator, within 72 hours prior to Screening or study vaccination.
2. Has had a positive COVID-19 test within the 90 days prior to Screening or study vaccination.
3. Current or planned participation in any other interventional clinical trial.
4. Participation in research involving any investigational product within 45 days prior to Screening or study vaccination.
5. Receipt of any approved or authorized products intended to prevent SARS-CoV-2 infection within 6 months prior to Screening or study vaccination.
6. Receipt of blood products or immunoglobulins within 60 days prior to Screening or study vaccination.
7. Received influenza vaccination within 14 days prior to Screening or study vaccination, or any other vaccine within 30 days prior to Screening or study vaccination.
8. Any significant autoimmune, immunodeficiency disease/condition, or auto inflammatory disorder (e.g., any known immunoglobulin A [IgA] deficiency, human immunodeficiency virus [HIV] infection, acquired immunodeficiency syndrome [AIDS])
9. Has current active hepatitis B or hepatitis C infection (based on self-reported medical history).
10. Has a peripheral arterial oxygen saturation (SpO2) level <92% at Screening, uncontrolled or severe asthma (e.g., more than 1 hospitalization for asthma exacerbation within the 12 months prior to Screening), or other uncontrolled or severe chronic lung disease or known bronchial hyper-reactivity to viruses that, in the opinion of the site investigator, would pose a health risk to the individual if enrolled.
11. Has known active tuberculosis.
12. Unstable non-cardiac illness (acute or chronic illness) requiring hospitalization or medical procedure during the 90 days prior to Screening or study vaccination, or cardiac condition (acute or chronic) requiring hospitalization or medical procedure (e.g., stenting, cardiac surgery, etc.) during the 1 year prior to Screening or study vaccination.
13. History of myocarditis, pericarditis, myopericarditis, or idiopathic cardiomyopathy, or presence of any medical condition (e.g., viral illness within 30 days of Screening or study vaccination) that, in the opinion of the investigator, increases risk of myocarditis, pericarditis, or myopericarditis.
14. Chronic kidney disease requiring dialysis or any type of ultrafiltration. Individuals with chronic kidney disease that does not require dialysis or ultrafiltration may be included.
15. Individuals with advanced or decompensated chronic liver disease as determined by the site investigator.
16. Presence of any transplanted solid organs (heart, kidney, lung, liver, pancreas, and/or intestine) or prior receipt of a blood stem cell transplant.
17. Administration of immunosuppressants, systemic glucocorticoids, or other immune-modifying drugs within the following timeframes:

    1. B-cell therapies within the 6 months prior to Screening or study vaccination.
    2. Prednisone, ≥20 mg or equivalent for more than 2 weeks, within the 30 days prior to Screening or study vaccination.
    3. Monoclonal antibodies that may suppress aspects of immune response (e.g., Dupixent) within the 6 months prior to Screening or study vaccination.
    4. Other medications in this category, including but not limited to high-dose inhaled corticosteroids (>800 mcg/day of beclomethasone dipropionate or equivalent); antimetabolites; transplant immunosuppressive agents; alkylating agents; cell-depleting agents; or cancer chemotherapeutics, within the 90 days prior to Screening or study vaccination.
    5. Any medication for any period of time that, in the opinion of the site investigator, could impede immune response to vaccination.
18. Known contraindication to IM injection (e.g., bleeding diathesis, acquired coagulopathy) or to IN administration (e.g., significant nasal abnormality or severe nasal obstruction, significant chronic rhinitis or history of chronic rhinitis, nasal septal defect causing significant breathing problems, unrepaired cleft palate, nasal polyps, or other nasal abnormality that might affect vaccine administration).
19. Receipt or anticipated receipt, within 7 days prior through 7 days after study vaccination, of any Intranasal medication, including FDA-approved prescription or over-the-counter products or non-FDA-approved alternative medicine products (e.g., Ayurvedic oil or other naturopathic substances).
20. Anticipated use of nasal irrigation (e.g., Neti PotTM) from Screening through 30 days after study vaccination.
21. Any known allergies to components contained in NDV-HXP-S (including egg products) or the comparator vaccine (including polyethylene glycol [PEG] allergies).
22. Women who are pregnant, breastfeeding, or who plan to become pregnant during the study.
23. Current or prior potential for NDV exposure (e.g., prior NDV-based vaccination, NDV-based oncologic immunotherapy, prior or current experience as a bird-handler, poultry farmer, or scientist conducting research with NDV).
24. Individuals who will have close or household high-risk contacts, within 14 days following study vaccination, including but not limited to:
25. Any other condition that, in the opinion of the site investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the investigational product or interpretation of study results.
26. Study team member or first-degree relative of any study team member (inclusive of CastleVax and site personnel involved in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of the NDV-HXP-S-KP.2 Vaccine Compared With an Approved mRNA COVID-19 Vaccine | Up to 180 days after vaccination
  Safety and tolerability of the NDV-HXP-S-KP.2 vaccine given intranasally and an approved mRNA COVID-19 vaccine given intramuscularly will be assessed in previously immunized adults. Outcomes include the percentage of participants with solicited local and systemic reactogenicity symptoms through 7 days, unsolicited adverse events through 30 days, and serious, medically attended, or special interest adverse events through 180 days. Clinically significant abnormal lab results (chemistry and hematology) will also be assessed through 7 days post-vaccination.

SECONDARY OUTCOMES:
Percentage of Participants With Viral Vector-Related Illness or Shedding After Vaccination | Through Day 31 post-vaccination
  The percentage of participants who experience symptoms suggestive of viral vector-related illness at Days 2, 8, 14, and 31 after vaccination will be assessed. The percentage of participants who test positive for viral vector shedding on Day 1 and at Days 2, 8, 14, and 31 post-vaccination will also be evaluated. In addition, the study will monitor whether any household contacts of participants develop symptoms of potential viral vector-related illness at Days 2 and 8 after vaccination.
Humoral Immune Response to the NDV-HXP-S-KP.2 Vaccine Compared With the Comparator Vaccine | From Day 1 through Day 181 post-vaccination
  The humoral immune response to the NDV-HXP-S-KP.2 vaccine administered intranasally and the comparator vaccine administered intramuscularly in previously immunized adults will be assessed through Day 181 after vaccination. Measurements will include serum geometric mean titers (GMTs) of SARS-CoV-2-specific neutralizing antibodies at Day 1 and at Days 31, 91, and 181 post-vaccination; serum geometric mean fold rise (GMFR) of SARS-CoV-2-specific neutralizing antibodies relative to Day 1 at Days 31, 91, and 181; serum GMTs of spike (S) protein-specific immunoglobulin G (IgG) binding antibodies at Day 1 and at Days 31, 91, and 181; and serum GMFR of S protein-specific IgG binding antibodies relative to Day 1 at Days 31, 91, and 181 post-vaccination.
Mucosal Immune Response to the NDV-HXP-S-KP.2 Vaccine Compared With the Comparator Vaccine | From Day 1 through Day 181 post-vaccination
  The mucosal immune response to the NDV-HXP-S-KP.2 vaccine administered intranasally and the comparator vaccine administered intramuscularly in previously immunized adults will be assessed through Day 181 after vaccination. Measurements will include the nasal lining fluid (NLF) geometric mean titers (GMTs) of spike (S) protein-specific secretory immunoglobulin A (sIgA) binding antibodies and total sIgA at Day 1 and at Days 31, 91, and 181 post-vaccination, as well as the geometric mean fold rise (GMFR) of S protein-specific sIgA binding antibodies and total sIgA relative to Day 1 at Days 31, 91, and 181 post-vaccination.

OTHER OUTCOMES:
Percentage of Participants Who Test Positive for SARS-CoV-2 After Vaccination | From Day 15 through Day 181 post-vaccination
  The percentage of participants who are identified as SARS-CoV-2-positive at any time from Day 15 through Day 181 after vaccination will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Egan, PhD, Study Chair — CastleVax Inc.
Locations (2):
- United States (2):
  - Skylight Health Research, Colorado Springs, Colorado
  - Skylight Health Research, Burlington, Massachusetts

IPD SHARING:
Plan to Share IPD: No
IPD will only be used internally at CastleVax for evaluation of the study outcomes.